CLINICAL TRIAL: NCT00005963
Title: Phase II Trial of Docetaxel and Carboplatin as First-Line Therapy for Metastatic Breast Cancer
Brief Title: Docetaxel and Carboplatin in Treating Women With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N9932; CDR0000067945 (Registry Identifier: PDQ (Physician Data Query)); NCI-2012-02341 (Registry Identifier: CTRP (Clinical Trials Reporting System))
Record Dates: First submitted 2000-07-05; First posted 2003-12-23 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Carboplatin; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- docetaxel + carboplatin (Experimental): This is a multicenter study. Patients receive docetaxel IV over 1 hour and carboplatin IV over 30 minutes on day 1. Treatment repeats every 3 weeks in the absence of disease progression or unacceptable toxicity. Patients who achieve stable disease (SD), partial response (PR), or complete response (CR) may receive 4 additional courses past SD, PR, or CR. Patients are followed every 6 months for 2 years and then annually for 3 years.
  Interventions: Drug: carboplatin; Drug: docetaxel

INTERVENTIONS:
Drug: carboplatin
Drug: docetaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one chemotherapy drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining docetaxel and carboplatin in treating women who have metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the anti-tumor activity of docetaxel and carboplatin in women with metastatic adenocarcinoma of the breast. II. Determine the objective response rate, time to progression, and survival in patients treated with this regimen. III. Determine the toxic effects of this regimen in these patients. IV. Assess the common functional polymorphisms in genes involved in chemotherapeutic response to improve prediction of clinical outcomes and provide insight into the potential for genotype-specific drug dosage.

OUTLINE: This is a multicenter study. Patients receive docetaxel IV over 1 hour and carboplatin IV over 30 minutes on day 1. Treatment repeats every 3 weeks in the absence of disease progression or unacceptable toxicity. Patients who achieve stable disease (SD), partial response (PR), or complete response (CR) may receive 4 additional courses past SD, PR, or CR. Patients are followed every 6 months for 2 years and then annually for 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven metastatic adenocarcinoma of the breast Measurable disease At least 20 mm in at least 1 dimension Hormone receptor status: Not specified

PATIENT CHARACTERISTICS: Age: 18 and over Sex: Female Menopausal status: Not specified Performance status: ECOG 0-2 Life expectancy: At least 3 months Hematopoietic: Granulocyte count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than upper limit of normal (ULN) SGOT/SGPT no greater than 2.5 times ULN Alkaline phosphatase no greater than ULN OR SGOT/SGPT no greater than ULN Alkaline phosphatase no greater than 4 times ULN Renal: Creatinine no greater than 1.5 times ULN Cardiovascular: No myocardial infarction within the past 6 months No congestive heart failure No unstable angina No clinically significant pericardial effusion or arrhythmia Other: No other invasive malignancy within the past 5 years except curatively treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix No active unresolved infection No prior hypersensitivity reaction to docetaxel No grade 2 or greater sensory or motor neuropathy Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent prophylactic filgrastim (G-CSF) during the first course of study therapy Chemotherapy: No prior chemotherapy for metastatic disease Prior adjuvant chemotherapy allowed More than 1 year since prior paclitaxel, docetaxel, cisplatin, or carboplatin No other concurrent chemotherapy Endocrine therapy: Not specified Radiotherapy: At least 4 weeks since prior radiotherapy to breast, chest wall, or axilla No prior radiotherapy to greater than 30% of bone marrow No concurrent radiotherapy Surgery: At least 4 weeks since prior major surgery and recovered Other: More than 7 days since prior IV antibiotics No concurrent experimental drugs

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2000-11; Primary Completion 2002-10 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
objective response rate | Up to 5 years

SECONDARY OUTCOMES:
time to progression | Up to 5 years
survival | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Edith A. Perez, MD, Study Chair — Mayo Clinic
Locations (21):
- United States (21):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Ochsner, New Orleans, Louisiana
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Medcenter One Health System, Bismarck, North Dakota
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Altru Health Systems, Grand Forks, North Dakota
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - CCOP - Geisinger Clinic and Medical Center, Danville, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota

REFERENCES:
- [Result] Perez EA, Suman VJ, Fitch TR, Mailliard JA, Ingle JN, Cole JT, Veeder MH, Flynn PJ, Walsh DJ, Addo FK. A phase II trial of docetaxel and carboplatin as first-line chemotherapy for metastatic breast cancer: NCCTG study N9932. Oncology. 2005;69(2):117-21. doi: 10.1159/000087813. Epub 2005 Aug 23. PMID 16118507